CLINICAL TRIAL: NCT01751035
Title: Integrative Risk Reduction and Treatment for Teen Substance Use Problems and PTSD
Acronym: RRFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00009042; R01DA031285-01 (NIH)
Record Dates: First submitted 2012-11-15; First posted 2012-12-17 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: PTSD; Alcohol Use Disorders; Substance Use Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual (TAU) (Placebo Comparator): Treatment as Usual (TAU) will be defined as it already exists within the community child advocacy centers. This could include individual and/or group therapy using a variety of treatment models.
  Interventions: Behavioral: Treatment as Usual
- RRFT (Experimental): RRFT is an acronym for an experimental intervention named Risk Reduction through Family Therapy. Please see intervention description for more detail about the model.
  Interventions: Behavioral: Risk Reduction through Family Therapy

INTERVENTIONS:
Behavioral: Risk Reduction through Family Therapy — RRFT is an integrative, ecologically-based approach to risk reduction and treatment. A Stage 1a feasibility trial and a Stage 1b pilot randomized controlled trial (RCT) evaluating RRFT have been completed. This Stage 1 work has resulted in a treatment manual, a clinician training protocol, and a quality assurance system. Preliminary findings from these studies are promising, indicating that RRFT can be readily learned and implemented with fidelity, and that it can lead to improvements in drug use and drug use-related risk and protective factors, PTSD symptoms, and risky sexual behaviors.
  Other Names: RRFT
  Arms: RRFT
Behavioral: Treatment as Usual — Participants assigned to the TAU condition will receive the standard treatment that a CSA victim would typically receive at community advocacy centers. In addition to treatment that is typically offered at the CACs, this will include a referral for substance abuse evaluation and may include referrals to other agencies in the community. TAU has been utilized as a comparison condition for several behavioral treatment evaluations involving adolescent substance abuse.
  Other Names: TAU
  Arms: Treatment as Usual (TAU)

SUMMARY:
Adolescents receiving RRFT and their caregivers will report significantly fewer substance use problems (quantity of use, frequency of use, and abuse symptoms) during treatment and follow-up than control adolescents who receive Treatment as Usual (TAU). Adolescents receiving RRFT and their caregivers will report improvement in empirically-demonstrated risk and protective factors for substance use and abuse at the individual level (e.g., coping) and at each level of an adolescent's ecology (e.g., increased number of positive family activities, reduced family conflict, reduced number of peers who use drugs, improved school attendance, increased involvement in pro-social community activities) during treatment and follow-up than control adolescents who receive TAU. Adolescents receiving RRFT will experience less PTSD symptoms (per youth and caregiver reports) during treatment and follow-up than control adolescents who receive TAU. Adolescents receiving RRFT will report engaging in fewer risky sexual behaviors (e.g., increased condom use, fewer partners) during treatment and follow-up than control adolescents who receive TAU. Changes during treatment in family relations (familial cohesiveness and conflict, satisfaction with caregiver-youth relationship) and parenting practices (monitoring) will mediate changes in substance use. Changes during treatment in emotional reactivity will mediate changes in PTSD symptoms.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* 1) 13-18 years old;
* 2) Presenting to LCC/HH for evaluation or treatment;
* 3) Report having experienced IPV in their lifetime, including: CSA, defined as forced or unwanted: (a) vaginal or anal penetration by an object, finger, or penis; (b) oral sex; (c) touching of the respondent's breasts or genitalia; or (d) respondents' touching of another person's genitalia; CPA, defined as having been (a) attacked or threatened with a gun, knife, or some other weapon; (b) attacked by another person with perceived intent to kill or seriously injure; (c) beaten and injured (i.e., "hurt pretty badly") by another person; (d) spanked so forcefully that it resulted in sustained welts or bruises or required medical care; or (e) cut, burned, or tied up by a caregiver as a punitive consequence; Exposure to Domestic Violence; and being victim of or bearing witness to Community Violence.
* 4) Have a memory of the incident(s);
* 5) Five or more DSM-IV PTSD symptoms;
* 6) Substance use, defined as alcohol or illicit drug use in the past 90 days per self-report and/or urine drug screen or breathalyzer.

Exclusion Criteria:

* 1) Previously identified as having a Pervasive Developmental Disability or Moderate to Severe Mental Retardation;
* 2) Actively suicidal or homicidal;
* 3) Reports active psychotic disorder

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 135 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
change in substance use problems (initiation/continuation, quantity, and abuse symptoms) | 18 months

SECONDARY OUTCOMES:
change in PTSD severity and symptoms | 18 months
change in risky sexual behaviors | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Carla K Danielson, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Danielson CK, Adams Z, McCart MR, Chapman JE, Sheidow AJ, Walker J, Smalling A, de Arellano MA. Safety and Efficacy of Exposure-Based Risk Reduction Through Family Therapy for Co-occurring Substance Use Problems and Posttraumatic Stress Disorder Symptoms Among Adolescents: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Jun 1;77(6):574-586. doi: 10.1001/jamapsychiatry.2019.4803. PMID 32022827